CLINICAL TRIAL: NCT00492505
Title: A Phase II Pilot Trial of Sorafenib, Tamoxifen and Cisplatin as Adjuvant Therapy for Patients With Stage III Malignant Melanoma
Brief Title: Sorafenib, Tamoxifen, and Cisplatin in Treating Patients With High-Risk Stage III Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Diego Pacific Oncology & Hematology Associates (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000551556; POHA-0602
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-07

CONDITIONS: Melanoma (Skin)
Keywords: stage IIIA melanoma; stage IIIB melanoma; stage IIIC melanoma
MeSH Terms: conditions — Melanoma | interventions — Cisplatin; Sorafenib; Tamoxifen; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: cisplatin
Drug: sorafenib tosylate
Drug: tamoxifen citrate
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as tamoxifen and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with tamoxifen and cisplatin after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying the side effects and how well giving sorafenib together with tamoxifen and cisplatin works in treating patients with high-risk stage III melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare relapse-free and overall survival of patients with high-risk stage III melanoma receiving adjuvant sorafenib tosylate, tamoxifen citrate, and cisplatin vs historical data from patients treated with tamoxifen citrate and cisplatin.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a pilot study. Patients are stratified according to number of positive lymph nodes identified during surgery.

Patients receive oral sorafenib tosylate twice daily on days 1-28, oral tamoxifen citrate twice daily on days 1-7, and cisplatin IV over 1 hour on days 2 and 3. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for at least 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of melanoma

  * High-risk, stage III disease
* No measurable metastatic disease
* Has undergone surgery within the past 8 weeks

  * Surgically rendered disease free

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Creatinine clearance ≥ 50 mL/min OR creatinine ≤ 1.5 mg/dL
* Liver function tests ≤ 3 times the upper limit of normal
* ANC ≥ 1,200/mm³
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm³
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No myocardial infarction within the past 6 months
* No congestive heart failure requiring medication
* No pulmonary disease requiring supplemental oxygen
* No dyspnea at rest
* No active infection
* No chronic underlying immunodeficiency disease
* No other serious illness that, in the physicians' opinion, may compromise the safety of the patient
* No other cancer within the past 5 years except for nonmelanoma skin cancer and cervical cancer
* No thromboembolic disease within the past 6 months

PRIOR CONCURRENT THERAPY:

* No prior tamoxifen citrate, sorafenib tosylate, or cisplatin
* No concurrent radiotherapy or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-04; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival
Overall survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Edward F. McClay, MD, Principal Investigator — San Diego Pacific Oncology & Hematology Associates
Locations (1):
- San Diego Pacific Oncology and Hematology Associates, Incorporated - Encinitas, Encinitas, California, United States